CLINICAL TRIAL: NCT04591964
Title: Effects of Remote Monitoring of Patients With Heart Failure Based on Smartphone Application: Open-labled Randomized Clinical Trial.
Brief Title: Effects of Remote Monitoring of Patients With Heart Failure Based on Smartphone Application
Acronym: ERICA-HF
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Principal Investigator, Akmaral Rustambekovna, Researcher in department of Chronic Heart Failure, National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0007188
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: CHF
Keywords: Chronic heart failure; telemedicine; mobile health; mobile application; remote monitoring

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, open-labled, comparative, randomized clinical trial.
  Baseline group: standard medical treatment + using of mobile application for remote monitoring, base of self-controlling, 12 month.
  Control group: standard medical treatment + base of self-controlling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- baseline (Active Comparator): standard medical therapy + using of mobile application + improving therapy
  Interventions: Combination Product: mobile application "M-Cardio" based on android
- Control (No Intervention): standard medical therapy

INTERVENTIONS:
Combination Product: mobile application "M-Cardio" based on android — Mobile apllication "M-Cardio" (android) for remote monitoring of patients with CHF developed on algorithms of clinical indicators, that's give us to evaluate current condition of patient, depends from quantity points of abnormals higher or lower threshold values, with automatically notification for doctor and patient for timely medical service.
  Arms: baseline

SUMMARY:
CHF is a most wild-spread and prognostically poor outcome most of cardiovascular and other disease. Despite of significant progress in treatment of CHF for the last years, death from this pathology stayed very high, reaching 60% for men, 45% for women during the 5 years after establishing diagnosis. The purpose of treatment is creating "seamless" system of care the whole continuum stretch CHF, in this connection, the particular relevance take in creating of new way and strategy with IT-technology mHealth. On the whole, mHealth application potentially suggest economic efficiency solution with continuous access for symptoms monitoring, stimulation of patients to self-servicing, self-controlling and achieving better results compare with optimal medical therapy. So, remote monitoring of patients on the base of mobile application must improve clinical and economic efficiency of medical care received.

In trial will be studied efficiency of using mobile application for remote monitoring of patients with ischemic etiology HF, also quality of life, commitment to therapy and prognosis (frequency of cardiovascular poor outcomes). Clinical indicators and tests (Quality of Life Minnesota Living with Heart Failure Questionnaire, Hospital Anxiety and Depression Scale, 6-minute walking test) will be evaluated in the beginning of the trial and repeatly after 1 year.

Trial financed by Kyrgyz Republic Ministry of Education and Science.

DETAILED DESCRIPTION:
It is single-centered, open-labled, comparative, prospective, randomized clinical trial, intended to study the benefits, if that's have, 12-month remote monitoring with using mobile application based on chronic heart failure clinical flow of 200 patients with coronary heart disease.

Participants will seen twice: screening, initial randomization, last 12 month, during which will be evaluated clinical and laboratory indicators. At the time of first screening visit will be singed informed consent. In the department of chronic heart failure of National Center of Cardiology and Internal Medicine named by M. Mirrakhimov the patients will be laboratory and clinical-instrumentary examined and have been teaching for using mobile application, basics of self-servicing and self-controlling. Participants, meeting all inclusion criteria, will come back for randomization during the hospitalization or just to standard medical therapy, or to standard medical therapy and remote monitoring with mobile application. In active comparator patients besides of standard medical therapy will use mobile application twice a week, if necessary every day, also foreseen two-way feedback with the coordinating doctor and online chat on WhatsApp.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over (not older 70 y.o)
* Participant willing and able to give informed consent
* Documented Coronary artery disease (CAD): either angio-graphically documented CAD or a previous history of myocardial infarction/angina.
* Verified heart failure functional class III (Nt-proBNP levels, 6-min walking test).
* Receiving basic therapy for CAD and chronic heart failure (CHF).
* Able (in the investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Cognitive impairments.
* Unstable course of CAD.
* Acute heart failure or CHF decompensation.
* Malignancy (receiving active treatment) or other life threatening disease.
* Renal dysfunction (stage 3B or worse).
* Thyroid dysfunction.
* Pregnancy/lactating females.
* Any other reason considered inappropriate by a study physician.
* Participants who have participated in any other clinical trial within the previous 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 12 month
  fixation of reaching the primary endpoint All-cause death
Recurrent hospitalizations due to chronic heart failure decompensation and/or non-fatal acute coronary syndrome. | 12 month
  fixation of reaching the primary endpoint recurrent hospitalizations due to chronic heart failure decompensation and/or non-fatal acute coronary syndrome.

SECONDARY OUTCOMES:
Quality of Life assesed Minnesota LIVING WITH HEART FAILURE Questionnaire (MLHFQ) | 12 month
  The questionnaire is comprised of 21 questions around several physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 (five) scale to indicate the extent to which each itemized adversity of heart failure has prevented the patient from living as they wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
  This questionnaire can be used as a key outcome measure in studies and evaluations of outpatients with symptomatic (NYHA class II to IV) heart failure with a reduced or preserved ejection fraction. This patient-reported outcome measurement tool can be used to determine whether a treatment for heart failure is effective for improving patients' quality of life by reducing the adverse impact of heart failure.
6-minute walking test results | 12 month
  The test is based on measuring the walking distance with turns along a long corridor (≥30 m) at the patient's own pace. Results will be evaluated at baseline and at 12 months
Nt-proBNP levels | 12 month
  Nt-proBNP levels will be evaluated while using mobile application for remote monitoring compared to lifestyle modification in patients with ischemic etiology CHF

OTHER OUTCOMES:
Сommitment | 12 month
  Will be assessed commitment of patients in baseline and control group using European Heart Failure Self-care Behaviour Scale (EHFScBS_9), which includes 9 items related to various issues of self-control. The responses are scaled from strongly agree - (1) to strongly disagree - (5). The total amount is calculated by adding up the points for each item. The lower the number of points reflects the better ability of patients with CHF for self-help.

CONTACTS AND LOCATIONS:
Overall Officials: Aigul Noruzbaeva, professor, Study Director — Head of CHF department
Locations (1):
- National Centre of Cardiology and Internal Medicine named after academician M.Mirrakhimov, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No